CLINICAL TRIAL: NCT04628247
Title: Effect of Spring Gravity Bar on Gait Pattern in Children With Spastic Diplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Baseem Zaki Mahmoud, BSc physiotherapy, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002557
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Spastic Diplegia Cerebral Palsy
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): They will receive the same traditional physical therapy exercise program in addition to gait training on spring gravity bar for one hour
  Interventions: Device: Spring gravity bar

INTERVENTIONS:
Device: Spring gravity bar — 1. contain two wooden board length (160 cm) and width (15 cm)
  2. contain pair of spring at every end of board
  3. two wooden board connect in the middle

SUMMARY:
The purpose of the study is to determine the effect of spring gravity bar on gait pattern in children with spastic diplegia

DETAILED DESCRIPTION:
The purpose of this study is to provide insight on investigate the effectiveness of vestibular stimulation on gait pattern by using spring gravity bar , when you bounce up and down it stimulate vestibular system that is considered straight line vestibular stimulation and strength extensor muscle of lower limb by pressure on spring during stance phase all that change gait stability and stride length so can improve gait pattern .

ELIGIBILITY:
Inclusion Criteria:

1. Their age will be extended from 7 to 10 years.
2. They can walk with limitation or holding on according to GMFCS (level II & II).
3. They can understand and follow instruction.

Exclusion Criteria:

- 1-children with any visual or auditory abnormalities. 2-children receiving any special medication affecting muscle and /or mental function.

3-children had any recent surgical interference in the lower limb. 4-children with perceptual defects. 5-children with fixed structural deformities lower limb.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Two dimensional gait analysis | 20 minute
  Two-dimensional (2D) video analysis may provide an accessible and affordable means of quantifying postural control deficits that can be implemented across a spectrum of care settings. Angular joint measures during weight lifting obtained using 2D motion analysis software have been shown to be highly correlated to goniometric measures . This system has also been shown to be reliable in quantifying range of motion during reaching and walking/running tasks
Dynamic gait index | 20 minute
  The Dynamic Gait Index is a sensitive and efficient tool for adults and therefore may be a useful tool for children. Dynamic Gait Index (DGI) is a performance-based tool that quantifiesthe dynamic balance instability developed by Shumway-Cook and Woollacott, evaluates the ability of the individual to modify gait in response to changing functions during walking

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Pediatric Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided